CLINICAL TRIAL: NCT03971786
Title: Sperm Parameters and Sexual Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A02455-50; 2018-53 (Other: Assistance Publique hopitaux de Marseille)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Men Infertility
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Quality of life — Assessment of quality of life through measuring scales

SUMMARY:
Infertility has important repercussions for couples in their emotional and sexual lives; the same is true of Assisted Procreation, which has an impact on the daily life of couples and a cost to society. Thus, fertility disorders are frequently associated with sexual dysfunction in both women and men (Khademi et al., 2008). In couples with male infertility, men have higher sexual dysfunction scores than couples with infertility without male aetiology (Smith et al., 2009).

To study the evolution of the sexual quality of life of infertile men before and after knowing their spermatic parameters

ELIGIBILITY:
Inclusion Criteria:

* Male patient presenting infertility status

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Variability of quality of life scoring with Male Sexual Health scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido, Study Director — Assistance Publique Hopitaux De Marseille

IPD SHARING:
Plan to Share IPD: No